CLINICAL TRIAL: NCT04476017
Title: An Open-Label Evaluation of the Safety and Tolerability of SAGE-718 in Participants With Parkinson's Disease Mild Cognitive Impairment
Brief Title: A Study to Evaluate the Safety and Tolerability of SAGE-718 in Participants With Parkinson's Disease Mild Cognitive Impairment (PD-MCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 718-CNP-201
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease; Cognitive Dysfunction
Keywords: Parkinson's Disease; Cognitive Dysfunction; SAGE-718
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The study had two parts: Part A and Part B with unique participants for each study part. Part B was started after Part A was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: SAGE-718 3 mg (Experimental): Participants received SAGE-718 3 milligrams (mg) tablets, once daily with food in the morning for 14 days.
  Interventions: Drug: SAGE-718
- Part B: SAGE-718 3 mg (Experimental): Participants received SAGE-718 3 mg tablets, once daily with food in the morning for 28 days.
  Interventions: Drug: SAGE-718

INTERVENTIONS:
Drug: SAGE-718 — Oral tablets.

SUMMARY:
The primary purpose of this two-part study was to evaluate the safety and tolerability of SAGE-718 and its effects on cognitive, neuropsychiatric, and motor symptoms in participants with Parkinson's disease mild cognitive impairment (PD-MCI).

ELIGIBILITY:
Inclusion Criteria:

1. Meet the following criteria for PD-MCI: Have a confirmed diagnosis of idiopathic PD according to 2015 Movement Disorder Society (MDS) clinical diagnostic criteria; Meet MDS Task Force Criteria for MCI in PD.
2. Have a score of 20 to 25 (inclusive) on the Montreal Cognitive Assessment (MoCA) at Screening.
3. Meet criteria for Hoehn & Yahr Stage I to III (mild to moderate motor severity) at Screening.
4. Have stable motor symptoms for at least 4 weeks prior to screening, in the opinion of the investigator.

Exclusion Criteria:

1. Have a diagnosis of dementia of any etiology, including but not limited to: Dementia associated with PD (probable or possible), Dementia with Lewy Bodies, Alzheimer's Dementia, and Vascular Dementia.
2. Have any indication of parkinsonism other than idiopathic PD.
3. In the opinion of the investigator, be experiencing unpredictable fluctuations in motor and/or nonmotor symptoms associated with PD.
4. Have an ongoing central nervous system condition other than idiopathic PD, including active neurologic and/or nonremitted psychiatric disorders, in the opinion of the investigator.
5. Have a history of brain surgery, deep brain stimulation, a significant head injury causing loss of consciousness greater than 30 minutes, or hospitalization due to a brain injury.
6. Have experienced significant psychotic symptoms within the past 3 months, including those associated with PD medications, as determined by the investigator.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Sage Investigational Site, Long Beach, California
  - Sage Investigational Site, Port Charlotte, Florida
  - Sage Investigational Site, West Palm Beach, Florida
  - Sage Investigational Site, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 4 investigative sites in the United States and took part in the study that ran from 31 July 2020 to 25 March 2022.
Groups:
- Part A: SAGE-718 3 mg: Participants received SAGE-718 3 milligrams (mg) tablets, once daily with food in the morning for 14 days in Part A of study.
- Part B: SAGE-718 3 mg: Participants received SAGE-718 3 mg tablets, once daily with food in the morning for 28 days in Part B of study.
Period: Part A (28 Days)
Arm/Group | Part A: SAGE-718 3 mg | Part B: SAGE-718 3 mg
Started | 11 | 0
Completed | 10 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Part B (42 Days)
Arm/Group | Part A: SAGE-718 3 mg | Part B: SAGE-718 3 mg
Started (Part B of this study was started after completion of Part A. Participants who completed Part A of the study were not included in Part B of the study. Unique participants were enrolled in Part B.) | 0 | 7
Completed | 0 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were administered investigational product (IP).
Groups:
- Part A: SAGE-718 3 mg: Participants received SAGE-718 3 mg tablets, once daily with food in the morning for 14 days in Part A of study.
- Total: Total of all reporting groups
Arm/Group | Part A: SAGE-718 3 mg | Part B: SAGE-718 3 mg | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Continuous [Mean (Full Range); unit: years] | 69.1 [51 to 74] | 70.3 [63 to 75] | 69.6 [51 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 9 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 7 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 7 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered with a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an IP whether or not related to the product. An AE can include any undesirable medical condition, even if no study treatment has been administered. TEAEs were defined as an AE with an onset date on or after the date of the first dose of IP or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study. Percentages are rounded off to the nearest single decimal.
Time Frame: From first dose of study drug up to 28 days
Population: Safety Set included all participants who were administered IP.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-718 3 mg
Number analyzed (Participants) | 11
percentage of participants | 45.5

2. Primary Outcome: Part B: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An AE was any untoward medical occurrence in a participant administered with a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an IP whether or not related to the product. An AE can include any undesirable medical condition, even if no study treatment has been administered. TEAEs were defined as an AE with an onset date on or after the date of the first dose of IP or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study. Percentages are rounded off to the nearest single decimal.
Time Frame: From first dose of study drug up to 42 days
Population: Safety Set included all participants who were administered IP.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: SAGE-718 3 mg
Number analyzed (Participants) | 7
percentage of participants | 14.3

3. Secondary Outcome: Part A and B: Percentage of Participants With Clinically Significant Changes in Vital Sign Measurements
Description: Vital signs included temperature, respiratory rate, heart rate (supine and standing), systolic blood pressure (supine and standing) and diastolic blood pressure (supine and standing). Percentage of participants with clinically significant change in vital signs measurements which were deemed clinically significant by the investigator were reported.
Time Frame: From first dose of study drug up to 28 days for Part A, and up to 42 days for Part B
Population: Safety Set included all participants who were administered IP.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-718 3 mg | Part B: SAGE-718 3 mg
Number analyzed (Participants) | 11 | 7
percentage of participants | 0 | 0

4. Secondary Outcome: Part A and B: Percentage of Participants With Clinically Significant Changes in Laboratory Assessments
Description: Laboratory tests assessments included hematology, biochemistry, coagulation and urinalysis. Percentage of participants with clinically significant change in laboratory assessments which were deemed clinically significant by the investigator were reported.
Time Frame: From first dose of study drug up to 28 days for Part A, and up to 42 days for Part B
Population: Safety Set included all participants who were administered IP.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-718 3 mg | Part B: SAGE-718 3 mg
Number analyzed (Participants) | 11 | 7
percentage of participants | 0 | 0

5. Secondary Outcome: Part A and B: Percentage of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Measurements
Description: Supine 12-lead ECGs were performed in triplicate and the standard intervals (heart rate, PR interval, QRS duration, QT interval, and corrected QT interval by Fridericia [QTcF]). Percentage of participants with clinically significant change in ECG measurements which were deemed clinically significant by the investigator were reported.
Time Frame: From first dose of study drug up to 28 days for Part A, and up to 42 days for Part B
Population: Safety Set included all participants who were administered IP.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-718 3 mg | Part B: SAGE-718 3 mg
Number analyzed (Participants) | 11 | 7
percentage of participants | 0 | 0

6. Secondary Outcome: Part A and B: Percentage of Participants With a Response of 'Yes' to Any Suicidal Ideation or Suicidal Behaviors Item Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS scale consisted of a baseline evaluation (at screening) that assessed the lifetime experience of participants with suicidal ideation (SI) and suicidal behavior (SB) and a postbaseline evaluation that focused on suicidality since the last study visit. The C-SSRS included "yes" or "no"' responses for assessment of suicidal ideation and behavior as well as numeric ratings for the severity of ideation, if present (from 1 to 5, with 5 being the most severe). The C-SSRS SI items involved wish to be dead, non-specific active suicidal thoughts, active SI with any methods, active SI with some intent and active SI with a specific plan. The C-SSRS SB items involved preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt (non-fatal) and completed suicide. Percentage of participants with a response of 'yes' are reported for both suicidal ideation and behavior in this OM.
Time Frame: From first dose of study drug up to 28 days for Part A, and up to 42 days for Part B
Population: Safety Set included all participants who were administered IP.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-718 3 mg | Part B: SAGE-718 3 mg
Number analyzed (Participants) | 11 | 7
percentage of participants
  Suicidal Ideation | 0 | 0
  Suicidal Behavior | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days for Part A, and up to 42 days for Part B
Description: Safety Set included all participants who were administered IP.
Arm/Group | Part A: SAGE-718 3 mg | Part B: SAGE-718 3 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/7
Other Adverse Events (participants affected / at risk) | 5/11 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SAGE-718 3 mg (N=11) | Part B: SAGE-718 3 mg (N=7)
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Eye contusions (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
International normalized ratio increased (Investigations) | 1 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT04476017/Prot_002.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT04476017/SAP_001.pdf